CLINICAL TRIAL: NCT02130323
Title: Phase 3 Randomized Controlled Trial of Non-inferiority of Topical Imiquimod vs. LEEP for Women With Carcinoma In-situ of the Cervix
Brief Title: Topical Imiquimod vs. LEEP for Women With Carcinoma In-situ of the Cervix
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMCSD.2014.0040
Record Dates: First submitted 2014-04-24; First posted 2014-05-05 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical intraepithelial neoplasia, Imiquimod
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Loop Electrosurgical Excision Procedure (Active Comparator): Excision of the cervical transformation zone by way of the loop electrosurgical excision procedure (LEEP) or cold knife conization (CKC).
  Interventions: Procedure: Loop Electrosurgical Excision Procedure
- Imiquimod (Experimental): Imiquimod 12.5mg intravaginally once weekly for 16 weeks
  Interventions: Drug: Imiquimod

INTERVENTIONS:
Drug: Imiquimod — 12.5mg (5%) once a week vaginally for 16 weeks
  Other Names: Aldara
  Arms: Imiquimod
Procedure: Loop Electrosurgical Excision Procedure — Patients with CIN 2-3 will be randomized to receive intervention, CKC or LEEP versus medical therapy with Imiquimod.
  Other Names: LEEP
  Arms: Loop Electrosurgical Excision Procedure

SUMMARY:
OBJECTIVE: The standard of care for high grade cervical intraepithelial neoplasia grade 2 to 3 (CIN 2-3) has been the excision of the cervical transformation zone by way of a loop electrosurgical excision procedure (LEEP) or cold knife conization (CKC). However, it has been recognized that these procedures can increase the risks for pre-term labor in women who still desire to conceive. Recent studies have shown that medical treatment with Imiquimod, a topical immune response modulator, has significant effects on histological regression of CIN 2-3 when compared with placebo. The investigators propose that treatment with Imiquimod may be preferable offering similar outcomes on histological regression when compared with excision or ablation while potentially avoiding or reducing the number of surgical procedure that places them at risk for future pregnancies.

DETAILED DESCRIPTION:
MATERIALS AND METHODS: A randomized controlled trial of patients with CIN 2-3 to receive either surgical excision with LEEP or CKC versus medical therapy with Imiquimod once weekly inserted vaginally for 16 weeks. Inclusion criteria are women age 21 years or older with confirmed histological diagnosis of CIN 2-3 with a normal endocervical curettage (ECC) if obtained and satisfactory colposcopy (the transformation zone of the cervix was completely visualized.) Exclusion criteria include positive CIN2-3 on ECC, presence of cancer, pregnancy or lactation, immune deficiency, hepatitis, or hypersensitivity to Imiquimod. Patients will be randomized to receive excision with LEEP/CKC or Imiquimod 250 mg (5%) cream (12.5 mg of active ingredient) inserted vaginally once a week for 16 weeks.

The primary outcome will be histological regression to CIN 1 or less. Secondary outcomes will be complete histological regression, high-risk Human Papilloma Virus (HPV) clearance, Clearance of HPV 16, 18/45, and patient tolerance of Imiquimod regimen. Follow up with repeat pap, HPV typing to include 16 and 18/45 subtyping, and colposcopy with directed cervical biopsy will be performed at 6 months post initiation of treatment. Patients unable to complete at least 8 treatments and miss two treatments consecutively will be considered failures and offered immediate LEEP. Those patients that complete 8 treatments of Imiquimod will be reevaluated 6 months from initiating treatment. Demographic information will be obtained to include age, gravidity and parity, smoking history, and contraceptive use.

Descriptive statistics will include numbers and rates of occurrence with confidence intervals of regression, pre, and post-treatment HPV including HPV 16 and 18/45 typing, and adverse effects. The assumed regression rate for the LEEP arm varies within studies. We are choosing a conservative estimate of 85% regression rate from CIN2+ to CIN1 or less. More recently in a 2014 publication in the Journal of Virology (Author Antonio Frega, Journal of Clinical Virology 60 (2014) 39-43) 13% of the LEEP patients out of 475 had residual disease after LEEP. In this study they excluded the 10% of patients that had had positive margins on their LEEP specimen. We are not excluding them as this is intent to treat study. For Imiquimod the Grimm study found a 73.3% regression rate with those treated with the active ingredient. A non-inferiority-type design for two proportions using differences is used in which the difference between treatments is defined as medical treatment being preferable if the regression rate is not more than 15% below that of the excisional treatment. Comparison of the regression rates of the two treatments will be made by a non-inferiority Fisher's exact test.

Required sample size was assessed using the PASS software of the NCSS statistical package. Using power = 0.80 and alpha = 0.05, a power analysis predicts the need for 68 patients per arm for 136. Post-treatment HPV rates will be compared similarly. We will recruit 75 patients to each arm to buffer for a dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women older than age 21, military or civilian
* Negative pregnancy test results
* Confirmed CIN 2-3 on cervical biopsy with a negative endocervical curettage (ECC) and satisfactory colposcopy visualizing the complete transformation zone of the cervix.
* The patient will be available and in the San Diego area for 6 months after enrollment to complete the clinic visits and follow up.

Exclusion Criteria:

* Positive CIN 2-3 on ECC
* Presence of cancer
* Pregnancy or lactation
* Immuno-compromised (systemic lupus erythematosus, kidney transplant)
* Hepatitis
* Hypersensitivity to Imiquimod
* Ulcerative colitis
* Crohn's disease
* Human Immunodeficiency virus

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12-21 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Human Papillomavirus(HPV) Clearance | 6 months from treatment initiation
  HPV clearance will be determined by pathology and HPV testing, followed by colposcopy.
  Descriptive statistics will include numbers and rates of occurrence with confidence intervals of regression, pre and post-treatment HPV including Human Papillomavirus type 16 (HPV16) and HPV 18/45 typing, and adverse effects. A non-inferiority type design is used in which the difference between treatments is defined as medical treatment being preferable if the regression rate is not more than 10% below that of the excisional treatment. Comparison of the regression rates of the two treatments will be made by a non-inferiority Fisher's exact test.

SECONDARY OUTCOMES:
Evidence of local or systemic side effects of Imiquimod cream | Every 4 weeks after initiation of Imiquimod Arm for 16 weeks
  Patients will be seen in dysplasia clinic at Naval Medical Center San Diego (NMCSD) every 4 weeks while in treatment to determine tolerability of the Imiquimod Arm. Patients with significant symptoms will be asked to delay using Imiquimod until symptoms resolve before resuming. Patients unable to complete at least 4 weeks of treatment (1 treatment per week), will be offered immediate LEEP or surveillance at the 6 month follow up.
Evidence of local or systemic side effects of Imiquimod cream | Daily after initiation of Imiquimod treatment Arm, up to 6 months after study initiation
  Patients will be provided a daily phone number to a qualified nurse regarding any symptoms experienced while on the Imiquimod arm of the study. Patients will be instructed to be evaluated in the Emergency Department after clinic hours if needed for up to 6 months after study initiation.
Number of Participants with Serious and Non-Serious Adverse Events | Up to 6 months after study initiation
  All reported Adverse Events will be captured on the Adverse Event report.

CONTACTS AND LOCATIONS:
Overall Officials: Addie N Alkhas, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No